CLINICAL TRIAL: NCT00140387
Title: Phase I/II Study of a Prime-Boost Schedule of Human GM-CSF Gene Transduced Irradiated Prostate Allogeneic Cancer Cell Vaccines (Allogeneic Prostate GVAX®) in Hormone-naïve Prostate Cancer Patients
Brief Title: Prime-Boost Dose Scheduling Trial for Human GM-CSF Gene Transduced Irradiated Prostate Allogeneic Cancer Cell Vaccines (Allogeneic Prostate GVAX®)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cell Genesys (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G-9802
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2005-09-01 (Estimated); Status verified 2005-08

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; GVAX; Metastatic; Vaccine; Allogeneic cells
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Neoplasm Metastasis

INTERVENTIONS:
Biological: Immunotherapy allogeneic GM-CSF secreting cellular vaccine

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of priming vaccinations, and subsequent boosting vaccinations with Human GM-CSF Gene Transduced Irradiated Prostate Allogeneic Cancer Cell Vaccines (Allogeneic Prostate GVAX®). Clinical observations and laboratory measurements will be monitored to evaluate safety and toxicity. Additionally, the antitumor effects of Allogeneic Prostate GVAX® on serum PSA levels will be evaluated and antitumor responses will be quantitated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adenocarcinoma prostate cancer
* No evidence of measurable metastatic disease
* An ECOG performance status of 0 or 1

Exclusion Criteria:

* Previous hormonal therapy of any type for prostate cancer
* Any previous chemotherapy, or prior investigational therapy for prostate cancer
* Prior Immunotherapy
* Prior treatment with gene therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 1999-05; Study Completion 2001-03